CLINICAL TRIAL: NCT02364817
Title: Impact of Attention Deficit/Hyperactivity Disorder on the Post-detoxification Alcohol Relapse Rate
Brief Title: ADHD: Gaps Between Patients With Alcohol-dependence and Impact on Relapse
Acronym: AGADIR
Status: Completed | Type: Observational
Sponsor: University Hospital, Lille (Other)
Collaborators: Institute for Scientific Research on Beverages (France) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2013_09; 2014-A00132-45 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Alcoholism; Attention Deficit Disorder With Hyperactivity
Keywords: Attention Deficit Disorder with Hyperactivity; Alcohol Dependence; Adults; Treatment outcome; Mental Health
MeSH Terms: conditions — Alcoholism; Attention Deficit Disorder with Hyperactivity; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post-Detox Cohort: All the patients included should meet Diagnostic and Statistical Manual 4th edition revised (DSM-IV-Tr) criteria for Alcohol Dependance. They are all recruited at the end of an inpatient alcohol detoxification process (see inclusion criteria).
  The initial screening is performed just before the end of hospitalization. The subsequent follow-up is 12 weeks-long. There is no drug for abstinence maintenance during the study. The psychosocial intervention is based on the BRENDA model.
  Interventions: Behavioral: cognitive and psychiatric assessment

INTERVENTIONS:
Behavioral: cognitive and psychiatric assessment — Administered at baseline:
  * Clinical Institute Withdrawal Assessment for Alcohol (CIWA-Ar)
  * hyperactivity : Adult ADHD Self-Report Scale (ASRS), Wenders-Utah Rating Scale (WURS), Diagnostic Interview for Adult ADHD 2nd edition (DIVA 2.0)
  * psychiatric history : Mini International Neuropsychiatric Interview 5th edition (MINI 5.0), Personality Disorder Questionnaire for the DSM-IV (PDQ-4)
  * cognitive functions : Frontal Assessment Battery (FAB), Montreal Cognitive Assessment (MoCA)
  * impulsivity : Barratt's Impulsiveness scale 11th edition (BIS-11)
  * alcohol consumption: alcohol - timeline follow-back (A-TLFB) ,administered at baseline (month before hospitalization), week 4 visit, week 6 visit, and week 12 visit.
  * administered at week 12: ASRS

SUMMARY:
Some recent studies have found that adult attention deficit - hyperactivity disorder (ADHD) was frequent among patients with alcohol-dependence. However, no investigation has ever addressed whether ADHD may impact the drinking outcome.

Moreover, most of the different aforementioned studies assessed ADHD using the ADHD self-report scale (ASRS). The ASRS is a screening questionnaire that is of limited diagnostic value, and the overrepresentation of high-score ASRS among patients with alcohol-dependence could be in part due to differential diagnoses such as antisocial or borderline personality disorders, executive function impairments, or isolated impulsiveness.

The study aims to evaluate "ADHD: Gaps between patients with Alcohol Dependence and Impact on early Relapse" (AGADIR). In AGADIR, subjects with alcohol-dependence are recruited at the end of a residential detoxification program. They are assessed for ADHD using the ASRS, but also with a standardized diagnostic tool, i.e., the Diagnostic Interview for ADHD in adults (DIVA 2.0). Potential differential diagnoses are screened during the baseline visit. The patients are followed-up during the 12 first post-detox weeks, through a standardized psychosocial treatment. ASRS is re-performed at the end of the follow-up.

ELIGIBILITY:
Inclusion Criteria:

* current DSM-IV-Tr criteria for alcohol-dependence
* current residential alcohol detoxification program

Non-inclusion Criteria:

* concurrent alcohol withdrawal symptoms, i.e., CIWA-Ar ≥ 10
* benzodiazepine diazepam-equivalent dose > 30 mg
* medical history of neurological impairment (excluding alcohol-induced cognitive disorders)
* guardianship or loss of liberty
* pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with alcohol-dependence who undergo a residential alcohol detoxification program
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Cumulated rate of alcohol relapse | 12 weeks
  Cumulated rate of alcohol relapse during the 12 weeks following the detoxification program

SECONDARY OUTCOMES:
Psychometric properties of the ASRS | 12 weeks
  Psychometric properties of the ASRS by comparison with the DIVA 2.0 and the screening of differential diagnoses
Multivariate analysis of the alcohol relapse | 12 weeks
  Multivariate analysis of the cumulated rate of alcohol relapse during the 12 weeks following the detoxification program

CONTACTS AND LOCATIONS:
Overall Officials: Renaud Jardri, MD, PhD, Principal Investigator — University Hospital of Lille (CHU Lille), France
Locations (3):
- France (3):
  - Ch Le Vinatier, Bron
  - Department of Addiction Medicine, Lille
  - Department of Addiction Medicine, Saint-Amand-les-Eaux

IPD SHARING:
Plan to Share IPD: No